CLINICAL TRIAL: NCT03537937
Title: Pragmatic Investigation of optimaL Oxygen Targets (PILOT) Trial
Brief Title: Pragmatic Investigation of optimaL Oxygen Targets Trial
Acronym: PILOT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Responsible Party: Principal Investigator, Matthew Semler, Assistant Professor of Medicine, Vanderbilt University Medical Center
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 171272
Record Dates: First submitted 2018-05-15; First posted 2018-05-25 (Actual); Results first posted 2023-09-25 (Actual); Last update posted 2023-09-25 (Actual); Status verified 2022-11

CONDITIONS: Respiratory Failure
MeSH Terms: conditions — Respiratory Insufficiency

STUDY DESIGN:
Intervention Model Description: In the PILOT trial, the entire study ICU will be assigned to a single SpO2 target (cluster-randomized) and the ICU will switch between lower, intermediate, and higher SpO2 targets every two months in a randomly generated sequence (cluster-crossover).
Who Masked: Outcomes Assessor
Masking Description: Observer bias will be minimized by use of objective endpoints collected in duplicate by [1] study personnel blinded to group assignment and [2] automated data extraction from the electronic health record.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Lower SpO2 Target (Active Comparator): During invasive mechanical ventilation in a study location, the fraction of inspired oxygen will be titrated to target an arterial oxygen saturation of 90% (range 88-92%).
  Interventions: Other: Lower SpO2 Target
- Intermediate SpO2 Target (Active Comparator): During invasive mechanical ventilation in a study location, the fraction of inspired oxygen will be titrated to target an arterial oxygen saturation of 94% (range 92-96%).
  Interventions: Other: Intermediate SpO2 Target
- Higher SpO2 Target (Active Comparator): During invasive mechanical ventilation in a study location, the fraction of inspired oxygen will be titrated to target an arterial oxygen saturation of 98% (range 96-100%).
  Interventions: Other: Higher SpO2 Target

INTERVENTIONS:
Other: Lower SpO2 Target — SpO2 target 90% (range 88-92%)
  Arms: Lower SpO2 Target
Other: Intermediate SpO2 Target — SpO2 target 94% (range 92-96%)
  Arms: Intermediate SpO2 Target
Other: Higher SpO2 Target — SpO2 target 98% (range 96-100%)
  Arms: Higher SpO2 Target

SUMMARY:
Mechanical ventilation of ICU patients universally involves titration of the fraction of inspired oxygen (FiO2) to maintain arterial oxygen saturation (SpO2). Despite decades of ICU practice, however, the optimal SpO2 target remains unknown. Current guidelines offer divergent recommendations as to the optimal SpO2 target. Therefore, we propose a 2,250-patient cluster-randomized cluster-crossover trial comparing a lower SpO2 target (90%; range 88-92%), an intermediate SpO2 target (94%; range 92-96%), and a higher SpO2 target (98%; range 96-100%) with regard to the outcome of days alive and free of invasive mechanical ventilation.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years
2. Receiving mechanical ventilation through an endotracheal tube or tracheostomy
3. Admitted to the study ICU or admission to the study ICU from the emergency department is planned

Exclusion Criteria:

1. Known pregnancy or beta hCG level greater than the laboratory upper limit of normal in a patient capable of becoming pregnant
2. Known to be a prisoner

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2541 (Actual)
Dates: Start 2018-07-01 (Actual); Primary Completion 2022-01-31 (Actual); Study Completion 2022-01-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Matthew W Semler, MD, Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: Yes
The NIH's guidelines for data sharing will serve as the model for the approach we will follow for the proposed investigation;
  http://grants.nih.gov/grants/policy/data_sharing/data_sharing_guidance.htm
  Even though the final dataset will be stripped of identifiers prior to release for sharing, the inherent link between the period in which the patient was admitted to the study ICU and group assignment in a cluster-crossover trial introduces a significant risk for deductive disclosure of subjects. Thus, we will make the data and associated documentation available to users only under a data sharing agreement that provides for: (1) a commitment to using the data only for research purposes and not to identify any individual participant; (2) a commitment to securing the data using appropriate computer technology; and (3) a commitment to destroying or returning the data after analyses are completed.
Supporting Information: Study Protocol, SAP, Analytic Code

REFERENCES:
- [Derived] Shapiro JC, Casey JD, Qian ET, Seitz KP, Wang L, Lloyd BD, Stollings JL, Freundlich RE, Self WH, Rice TW, Wanderer JP, Semler MW; Pragmatic Critical Care Research Group. Oxygen Targets for Mechanically Ventilated Adults with Sepsis: Secondary Analysis of the PILOT Trial. J Intensive Care Med. 2025 May;40(5):486-494. doi: 10.1177/08850666241299378. Epub 2025 Jan 9. PMID 39784122
- [Derived] Semler MW, Casey JD, Lloyd BD, Hastings PG, Hays MA, Stollings JL, Buell KG, Brems JH, Qian ET, Seitz KP, Wang L, Lindsell CJ, Freundlich RE, Wanderer JP, Han JH, Bernard GR, Self WH, Rice TW; PILOT Investigators and the Pragmatic Critical Care Research Group. Oxygen-Saturation Targets for Critically Ill Adults Receiving Mechanical Ventilation. N Engl J Med. 2022 Nov 10;387(19):1759-1769. doi: 10.1056/NEJMoa2208415. Epub 2022 Oct 24. PMID 36278971
- [Derived] Semler MW, Casey JD, Lloyd BD, Hastings PG, Hays M, Roth M, Stollings J, Brems J, Buell KG, Wang L, Lindsell CJ, Freundlich RE, Wanderer JP, Bernard GR, Self WH, Rice TW; PILOT Investigators and the Pragmatic Critical Care Research Group. Protocol and statistical analysis plan for the Pragmatic Investigation of optimaL Oxygen Targets (PILOT) clinical trial. BMJ Open. 2021 Oct 28;11(10):e052013. doi: 10.1136/bmjopen-2021-052013. PMID 34711597

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Lower SpO2 Target | Intermediate SpO2 Target | Higher SpO2 Target
Started | 808 | 859 | 874
Completed | 808 | 859 | 874
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Lower SpO2 Target | Intermediate SpO2 Target | Higher SpO2 Target | Total
Number analyzed (Participants) | 808 | 859 | 874 | 2541
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 57 [44 to 67] | 59 [47 to 68] | 59 [45 to 68] | 58 [45 to 68]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 361 | 385 | 409 | 1155
  Male | 447 | 474 | 465 | 1386
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 2 | 0 | 2
  Asian | 10 | 11 | 7 | 28
  Native Hawaiian or Other Pacific Islander | 0 | 2 | 2 | 4
  Black or African American | 121 | 140 | 136 | 397
  White | 649 | 666 | 695 | 2010
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 28 | 38 | 34 | 100
Overall Number of Participants [Count of Participants; unit: Participants] | 808 | 859 | 874 | 2541
Overall Number of Participants [Count of Participants; unit: Participants] | 808 | 859 | 874 | 2541
Overall Number of Participants [Count of Participants; unit: Participants] | 808 | 859 | 874 | 2541

OUTCOME MEASURES:

1. Primary Outcome: Ventilator-free Days (VFDs) to Study Day 28
Description: Number of days alive and free from invasive mechanical ventilation between the final liberation from invasive mechanical ventilation before 28 days and study day 28. Patients who continue to receive invasive mechanical ventilation at day 28 or have died prior to day 28 will receive zero VFDs. For patients who return to invasive mechanical ventilation and are subsequently liberated from invasive mechanical ventilation prior to day 28, VFDs will be counted from final liberation from mechanical ventilation.
Time Frame: 28 days
Measure: Median (Inter-Quartile Range); unit: number of days
Arm/Group | Lower SpO2 Target | Intermediate SpO2 Target | Higher SpO2 Target
Number analyzed (Participants) | 808 | 859 | 874
number of days | 20 [0 to 25] | 21 [0 to 25] | 21 [0 to 26]

2. Secondary Outcome: 28-day, In-hospital Mortality (Secondary Outcome)
Description: All-cause mortality prior to discharge from the hospital, assessed at 28 days after enrollment (Secondary Outcome).
Time Frame: 28 days
Measure: Count of Participants; unit: Participants
Arm/Group | Lower SpO2 Target | Intermediate SpO2 Target | Higher SpO2 Target
Number analyzed (Participants) | 808 | 859 | 874
Participants | 281 | 292 | 290

3. Secondary Outcome: Intensive Care Unit Mortality (Exploratory Clinical Outcome)
Description: All-cause mortality prior to transfer out of the intensive care unit
Time Frame: 28 days
Measure: Count of Participants; unit: Participants
Arm/Group | Lower SpO2 Target | Intermediate SpO2 Target | Higher SpO2 Target
Number analyzed (Participants) | 808 | 859 | 874
Participants | 244 | 259 | 249

4. Secondary Outcome: Vasopressor-free Days (Exploratory Clinical Outcome)
Description: Number of days alive and free from vasopressor receipt between the final receipt of vasopressors before 28 days and study day 28.
Time Frame: 28 days
Measure: Median (Inter-Quartile Range); unit: number of days
Arm/Group | Lower SpO2 Target | Intermediate SpO2 Target | Higher SpO2 Target
Number analyzed (Participants) | 808 | 859 | 874
number of days | 25 [0 to 28] | 25 [0 to 28] | 25 [0 to 28]

5. Secondary Outcome: Renal Replacement Therapy-free Days (Exploratory Clinical Outcome)
Description: Number of days alive and free from renal replacement therapy between the final receipt of renal replacement therapy before 28 days and study day 28
Time Frame: 28 days
Measure: Median (Inter-Quartile Range); unit: number of days
Arm/Group | Lower SpO2 Target | Intermediate SpO2 Target | Higher SpO2 Target
Number analyzed (Participants) | 808 | 859 | 874
number of days | 28 [0 to 28] | 28 [0 to 28] | 0 [0 to 28]

6. Secondary Outcome: Intensive Care Unit-free Days (Exploratory Clinical Outcome)
Description: Number of days alive and free from intensive care unit admission after the final transfer out of the intensive care unit before 28 days to study day 28
Time Frame: 28 days
Measure: Median (Inter-Quartile Range); unit: number of days
Arm/Group | Lower SpO2 Target | Intermediate SpO2 Target | Higher SpO2 Target
Number analyzed (Participants) | 808 | 859 | 874
number of days | 20 [0 to 24] | 19 [0 to 24] | 20 [0 to 24]

7. Secondary Outcome: Hospital-free Days (Exploratory Clinical Outcome)
Description: Number of days alive and free from hospital admission to study day 28
Time Frame: 28 days
Measure: Median (Inter-Quartile Range); unit: number of days
Arm/Group | Lower SpO2 Target | Intermediate SpO2 Target | Higher SpO2 Target
Number analyzed (Participants) | 808 | 859 | 874
number of days | 10 [0 to 20] | 10 [0 to 21] | 10 [0 to 20]

8. Secondary Outcome: Acute Kidney Injury (AKI) (Exploratory Organ Function Outcome)
Description: Presence of Stage II or greater AKI by Kidney Disease: Improving Global Outcomes (KDIGO) criteria
Time Frame: 28 days
Measure: Count of Participants; unit: Participants
Arm/Group | Lower SpO2 Target | Intermediate SpO2 Target | Higher SpO2 Target
Number analyzed (Participants) | 808 | 859 | 874
Participants | 230 | 253 | 251

9. Other Pre Specified Outcome: Atrial Arrhythmia (Exploratory Safety Outcome)
Description: Documented atrial arrhythmia
Time Frame: 28 days
Measure: Count of Participants; unit: Participants
Arm/Group | Lower SpO2 Target | Intermediate SpO2 Target | Higher SpO2 Target
Number analyzed (Participants) | 808 | 859 | 874
Participants | 64 | 100 | 95

10. Other Pre Specified Outcome: Ventricular Arrhythmia (Exploratory Safety Outcome)
Description: Documented ventricular arrhythmia
Time Frame: 28 days
Measure: Count of Participants; unit: Participants
Arm/Group | Lower SpO2 Target | Intermediate SpO2 Target | Higher SpO2 Target
Number analyzed (Participants) | 808 | 859 | 874
Participants | 20 | 21 | 20

11. Other Pre Specified Outcome: Cardiac Arrest (Exploratory Safety Outcome)
Description: Cardiac arrest with return of spontaneous circulation
Time Frame: 28 days
Measure: Count of Participants; unit: Participants
Arm/Group | Lower SpO2 Target | Intermediate SpO2 Target | Higher SpO2 Target
Number analyzed (Participants) | 808 | 859 | 874
Participants | 26 | 26 | 31

12. Other Pre Specified Outcome: Pneumothorax or Pneumomediastinum (Exploratory Safety Outcome)
Description: Pneumothorax or pneumomediastinum as defined by documentation in the electronic health record by treating clinicians or radiology of a pneumothorax on thoracic imaging or thoracic ultrasound.
Time Frame: 28 days
Measure: Count of Participants; unit: Participants
Arm/Group | Lower SpO2 Target | Intermediate SpO2 Target | Higher SpO2 Target
Number analyzed (Participants) | 808 | 859 | 874
Participants | 17 | 24 | 36

13. Other Pre Specified Outcome: Ischemic Stroke (Exploratory Safety Outcome)
Description: New ischemic stroke between enrollment and 28 days after enrollment as diagnosed by computed tomography, magnetic resonance imaging, or cerebral angiography.
Time Frame: 28 days
Measure: Count of Participants; unit: Participants
Arm/Group | Lower SpO2 Target | Intermediate SpO2 Target | Higher SpO2 Target
Number analyzed (Participants) | 808 | 859 | 874
Participants | 12 | 17 | 16

14. Other Pre Specified Outcome: Myocardial Infarction (Exploratory Safety Outcome)
Description: New myocardial infarction between enrollment and 28 days after enrollment, defined as detection of a rise in cardiac troponin values with at least one value above the 99th percentile and clinical evidence of acute myocardial ischemia.
Time Frame: 28 days
Measure: Count of Participants; unit: Participants
Arm/Group | Lower SpO2 Target | Intermediate SpO2 Target | Higher SpO2 Target
Number analyzed (Participants) | 808 | 859 | 874
Participants | 16 | 28 | 14

ADVERSE EVENTS:
Time Frame: enrollment to day 28
Arm/Group | Lower SpO2 Target | Intermediate SpO2 Target | Higher SpO2 Target
All-Cause Mortality (participants affected / at risk) | 285/808 | 296/859 | 297/874
Serious Adverse Events (participants affected / at risk) | 0/808 | 0/859 | 0/874
Other Adverse Events (participants affected / at risk) | 1/808 | 0/859 | 0/874
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lower SpO2 Target (N=808) | Intermediate SpO2 Target (N=859) | Higher SpO2 Target (N=874)
Relative bradycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-06-10): https://cdn.clinicaltrials.gov/large-docs/37/NCT03537937/Prot_SAP_000.pdf